CLINICAL TRIAL: NCT05742282
Title: Validation of the AUB-HAS2 Score in a Brazilian Population and Study of the Additional Impact of Biomarkers in Predicting Perioperative Risk
Brief Title: ASPIRE (Aub-haS2 Plus bIomaRkErs)
Acronym: ASPIRE
Status: Not yet recruiting | Type: Observational
Sponsor: Hospital Samaritano Paulista (Other)
Responsible Party: Principal Investigator, Pedro Gabriel Melo de Barros e Silva, Director of Clinical Research, Hospital Samaritano Paulista
Other Study IDs: 001/23
Record Dates: First submitted 2023-02-11; First posted 2023-02-23 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Perioperative Medicine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
ASPIRE is a prospective, multicenter, observational study that will assess the performance of AUB-HAS2 to predict the occurrence of major adverse cardiovascular events 30-days after a non-cardiac surgery and the additional role of high-sensitivity troponin T and NT-ProBNP biomarkers in the accuracy of different event prediction indexes after non-cardiac procedures.

DETAILED DESCRIPTION:
Primary objectives:

Primary objective of the validation arm: to analyze the accuracy of the AUB-HAS2 index in predicting the occurrence of myocardial infarction, stroke and death within 30 days after non-cardiac surgeries.

Primary objective biomarker arm: to analyze the additional role of high-sensitivity troponin T and NT-ProBNP biomarkers in the accuracy of different event prediction indexes after non-cardiac surgeries.

Secondary objectives:

To analyze the potentially preventable factors related to adverse outcomes after non-cardiac surgeries in order to offer subsidies for more assertive guidelines regarding the implementation of perioperative protection strategies. Compare the performance of these scores with others that have already been validated (ACP and Lee - see Annex A).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 40 years, in the preoperative period of non-cardiac procedures, with expected hospitalization for at least 24 hours postoperatively.

Exclusion Criteria:

* Refusal to sign the informed consent form.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients ≥ 40 years, that will undergo non-cardiac procedures, with expected hospitalization for at least 24 hours postoperatively.
Sampling Method: Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 2025-06-21 (Estimated); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-10-30 (Estimated)

PRIMARY OUTCOMES:
RATE OF MAJOR ADVERSE CARDIOVASCULAR EVENTS | 30 days
  COMPOSITE OF DEATH, MYOCARDIAL INFARCTION AND STROKE

SECONDARY OUTCOMES:
RATE OF MYOCARDIAL INJURY | 30 days

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Samaritano Paulista, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided
Data can be shared under formal requisition and justification